CLINICAL TRIAL: NCT00547118
Title: The Effects of the Cannabinoid-1 Receptor Antagonist, Rimonabant, on Weight and Metabolic Risk Factors in People With Schizophrenia
Brief Title: The Effects of Rimonabant, on Weight and Metabolic Risk Factors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn due to medication withdrawal from the EMEA
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, MPRC, Robert Buchanan, MD, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00041206
Record Dates: First submitted 2007-10-19; First posted 2007-10-22 (Estimated); Results first posted 2015-02-27 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Obesity; Hypertension; Smoking
Keywords: Metabolic abnormalities; Safety; Satiety
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Obesity; Hypertension; Smoking | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Rimonabant
  Interventions: Drug: Rimonabant
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rimonabant — One 20 mg tablet given 1 time per day for 112 days.
  Arms: 1
Drug: Placebo — One placebo tablet given 1 time per day for 112 days.
  Arms: 2

SUMMARY:
1) To examine the efficacy of rimonabant in decreasing weight and metabolic parameters/cardiovascular disease risk in people with schizophrenia receiving second generation antipsychotics 2) To examine the safety and tolerability of rimonabant as an adjunctive agent for decreasing weight and metabolic risk in people with schizophrenia 3) To examine the efficacy of rimonabant for neurocognitive impairments in people with schizophrenia treated with second-generation antipsychotics (secondary outcome) 4) To examine the efficacy of rimonabant for patient perceived health outcomes and quality of life (secondary outcome) 5) To test the effect of rimonabant on cigarette smoking, nicotine dependence and nicotine craving in people with schizophrenia 6) To examine the effects of rimonabant on food satiety in people with schizophrenia

There is an increasing awareness of the problem of metabolic issues in people with schizophrenia and renewed focus on physical health care for this population. There is under-treatment, in general, of medical conditions in people with schizophrenia, and increased mortality from natural causes. People with schizophrenia are at risk for developing obesity due to many factors including inactive lifestyle, poor dietary choices, and side effects of the commonly used atypical antipsychotics. Metabolic syndrome has been discussed in the cardiology and endocrinology for over two decades, but its prevalence in the mentally ill is only now being fully realized. Diabetes mellitus may be twice as prevalent among patients with schizophrenia as in the general population and metabolic syndrome is probably even more prevalent than diabetes among people with schizophrenia. There is now an opportunity to address this serious problem. A new drug, rimonabant, has recently been approved in several European and Latin American countries. This drug represents the first of a new class of psychoactive drugs witch may improve metabolic problems through decreasing appetite drive. This may also help decrease the drive for cigarette use, which is also a great problem for people with schizophrenia. Is this a safe and effective treatment in this population? This study proposes to test this question in a rapid study, which will develop the basis for future work in this important area.

DETAILED DESCRIPTION:
Part I will be a 2-week evaluation phase. In Part I, subjects undergo a diagnostic interview for symptoms and treatment along with medical, side effect measures, and neuropsychological tests (tests for memory, attention, and motor task skills). An electrocardiogram (EKG), a urine sample, and about 3 tablespoons of blood will be taken for laboratory tests. Women will have a pregnancy test. This part of the study is 3-4 visits. The time of the visits will be about 8 hours.

Part II is a 16-week treatment phase subjects will be randomly assigned to either rimonabant or placebo for a 16-week period. The medication will be given in unmarked capsules so that subjects will not know which medication they are receiving. Only the pharmacist will know which medications subjects are receiving. If an emergency occurs we will break the blind and give appropriate care. This phase will require one visit every week and each visit may take up to 2-3 hours. Subjects will be examined every week to check symptoms side effects. Subjects symptoms will be evaluated using specially designed rating scales, to ask about their daily experiences and feelings. Evaluations that occur every 4 weeks may take about 2 hours. At week 8 and week 16 laboratory tests will be repeated. These tests will be compared to the baseline tests taken in Part I. The end of study tests may take up to a total of 8 hours and may require 3-4 visits. All testing is done for research purposes only and would not be performed if subjects were not participating in this study. The total number of visits requested for this study will be 16-20. When subjects undergo neuropsychological testing, we will examine their ability to learn and remember numbers and words to pay attention and to quickly perform motor tasks. A motor task is when you use your hands to perform a task such as placing pegs into a piece of wood. These tests will take about 2 hours and are done at the beginning of Part I and the end of Part II.

Diet and exercise counseling will be held weekly for groups and individuals. Sessions will focus on topics such as calories, fat content, portion control and determining a healthy weight. We will request that participants maintain a food diary and exercise approximately 30 minutes/3 times per week. Subjects will be encouraged to attend the counseling sessions. Transportation will be available for subjects. If patients have not attended sessions, they will be reeducated on the importance of attending sessions at the time of clinical ratings.Subjects will not be discharged from the study if they do not attend sessions.

Randomization will be done using a permuted block randomization system, and will be stratified by clozapine/olanzapine treatment at baseline. Treatment assignment order is random within each block, and the total number of patients assigned to each treatment is equal. The block sizes will vary between sizes 2 and 4 in random sequence. The unblinded pharmacist will be notified of the treatment assignment, and will inform unblinded pharmacists at the other sites about which study medication to dispense. In an emergency, research staff will be able to contact the pharmacy for unblinding. Rimonabant will be available in 20 mg capsules with matched placebo.

For outpatients study medication will be dispensed on a weekly basis plus two extra days of medication. Inpatient subjects will receive their study medication daily from the Maryland Psychiatric Research Center (MPRC) Treatment Research Program (TRP) central pharmacy by a non-blind pharmacist. The blind will be broken only if a medical emergency requires this information. If this occurs, the patient will be withdrawn from the study.

All raters, investigators and other staff will be blind to treatment assignment except for the pharmacist. The pharmacist does not participate in assessing any of the primary symptom or side effect dependent variables and conveys no information about treatment assignment to patients or staff except in a medical emergency.

Patients receiving 75% of their assigned medication will be considered compliant. Outpatient compliance will be monitored through weekly pill counts and subject interviews. Inpatient compliance will be monitored through inpatient medication records. If a patient is observed to be non-compliant then this will be discussed with the patient and a plan formulated to bring the patient back within the compliance parameter. For outpatients the plan may include contacting the patients caretaker or scheduling increased clinic visits. These monitoring procedures have been used in other MPRC studies and have resulted in high levels of compliance. Compliance patterns will be carefully monitored in each treatment group and will be described as part of any presentation of study results.

Satiety is defined as the reduced willingness to eat after a meal, not due to sickness or other extraneous factors and can be thought of as sensations of fullness. A preload and a test meal will be used in this study. The preload is a fixed amount of food given to the participant that is consumed in its entirety. The test meal is a food or foods served, following the preload, in sufficient quantity so that the participant can eat as much as desired. The amount consumed of the test meal is measured and used as an index of satiety. Likert and Visual Analog Scales (VAS) will also be used.

We will employ both the preload-test meal paradigm along with rating scales in the present study to investigate the effects of rimonabant on satiety signaling. The testing will occur at baseline, week 8, and week 16 to see if the effect changes. All three testing occasions will be the same. Participants will arrive after skipping breakfast and given a preload of 12 oz. of Ensure (375 kcal) served chilled in a large, plastic cup. Hunger ratings will be taken at baseline, then every 30 minutes for 90 minutes. After 60 minutes a test meal consisting of a pre-weighed bowl each of Reduced Fat Wheat Thins and Nilla Wafers will be given. These will be kept in separate bowls so that exact caloric consumption can be measured. The test meal will be served with 12 oz. of water served chilled in a large plastic cup. Satiety will be assessed by the quantity of Wheat Thins, Nilla Wafers, and water consumed and the difference between the hunger rating score from baseline for each time point.

About 75% of subjects will be smokers. Smoking measures will be performed on those with >8 ppm CO in expired breath and who smoke at least 5 cigarettes daily. One approach to studying tobacco craving in the laboratory is to compare smokers responses when exposed to neutral and smoking-related in vivo cues. In vivo or "real-life" cues are either presented by the experimenter or involve manipulation of materials by the participant. For this study, after smoking a cigarette at baseline (15 minutes before testing begins), patients will be asked to complete the Tobacco Craving Questionnaire (TCQ) and the Positive and Negative Affect Schedule (PANAS). Participants will then be exposed to two experimental trials presented in random order: 1) smoking cues, and 2) neutral cues.Each trial will last 20 minutes. Participants will complete the TCQ and PANAS immediately and 10 and 20 minutes after cue exposure. There will be a rest period between trials. During the rest period, the patient will complete other study assessments lasting 30-60 minutes. After the assessments, the patient will smoke again and then will complete the ratings and cue reactivity session for the second random condition at the same time points (baseline, immediately after, 10 and 20 minutes).Trials will begin with the experimenter placing a tray containing an opaque cover on a table in front of the participant. In the smoking cue condition, a pack of the participants preferred brand of cigarettes a lighter and an ashtray will be under the tray cover. In the neutral cue condition, a pack of unsharpened pencils and a pencil sharpener will be under the cover. When instructed, the participant will lift the cover on the tray. In the smoking cue condition, participants will take one cigarette out of the pack light it without puffing hold it and look at it. At the end of the exposure period participants will extinguish the cigarette, and replace the cover on the tray. In the neutral cue condition, participants will take one pencil out of the pack sharpen it hold it and look at it.

The Iowa Gambling Task (IGT) is a computer-administered cognitive test that measures risk-reward decision-making. Performance is impaired in patients with brain lesions in the ventromedial prefrontal cortex and in people who abuse alcohol, cocaine, marijuana, methamphetamine, opiates, or multiple illegal drugs. Patients with schizophrenia show normal IGT performance in some studies. In particular, adolescent patients and adults with catatonic schizophrenia show impairment. One study found that IGT performance was significantly correlated with negative symptoms. In this study, subjects will take one of two equivalent versions of the IGT at study entry and study completion. Each task session will take up to 30 minutes.

The Tobacco Craving Questionnaire (TCQ) is a questionnaire designed to assess current tobacco craving. Factor analysis of the 47-item TCQ resulted in four factors: 1) emotionality, smoking in anticipation of relief from withdrawal or negative mood; 2) expectancy, anticipation of positive outcomes from smoking; 3) compulsivity, an inability to control tobacco use; and 4) purposefulness, intention and planning to smoke for positive outcomes. We will use a 12-item version of the TCQ, comprising the three items from each factor that exhibited optimal within-factor reliability (Cronbachs coefficient alpha) and inter-item correlation. The 12-item TCQ is as valid and reliable as the 47-item version. TCQ items are rated on a scale from 1 strongly disagree to 7 strongly agre. Factor scale scores for each participant are obtained by summing the three items.

The PANAS is a 20-item scale in which 10 items describe positive mood (enthusiastic, interested, determined, excited, inspired, alert, active, strong, proud, attentive) and 10 items describe negative mood (scared, afraid, upset, distressed, jittery, nervous, ashamed, guilty, irritable, hostile). Each item is rated on a 5-point scale (not at all, a little, moderately, quite a bit, extremely). The PANAS shows high internal consistency and test-retest reliability. Subjects can leave the study at any point. If a participant experiences worsening of psychotic symptoms (relative to the baseline BPRS, an increase of 3 points or more OR an increase from a 5 to 7 on any one of the following BPRS items: somatic concern, conceptual disorganization, hostility, suspiciousness, hallucinatory behavior, or unusual thought content OR an increase of 2 or more on the CGI global severity OR the subject is judged to be entering an exacerbation of his/her illness by the treating clinician), the patient will be discontinued from the study. Other reasons for study termination include evidence of suicidal thinking or behavior, or the development of or worsening of significant depressive symptoms (score at any point in the study of >10 on the CDS or a 3 on the suicidal item), complete cessation of eating and drinking for > 24 hours, pregnancy, or blood pressure > 165/95 on three consecutive readings. Once a participant is discontinued from the study for whatever reason, completion ratings will be performed. This includes laboratory tests rating scales and neurocognitive assessments.

If a patient is prematurely terminated from the study, they will resume their standard treatment. At the end of the study patients will not have the option of continuing rimonabant because it is not FDA approved in the US. Other interventions to improve weight and metabolic profiles will be discussed with the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Any gender
2. Any race,
3. Age range of 18-55.
4. Meet DSM-IV (APA, 1994) criteria for either schizophrenia or schizoaffective disorder.
5. Have a BMI greater than or equal to 27 with treated or untreated hyperlipidemia/ hypertriglyceridemia or a BMI greater than or equal to 30 regardless of concurrent risk factors
6. Be treated with the same SGA for at least 8 weeks and to have received a constant therapeutic dose for at least 30 days
7. Be clinically stable (for inpatients: at least one month post admission). Hyperlipidemia and hypertriglyceridemia are defined by ATP III guidelines such that borderline high and high will be considered as criteria for these disorders (ATP III 2001).

Exclusion Criteria:

1. Subjects with significant recent depressive symptoms will be excluded from the study, defined as any history of a suicide attempt or suicidal ideation or hospitalization for depressive symptoms within the last 6 months; or a high level of current depressive symptoms (Calgary Depression Scale of > 7) (Addington 1993, Kim et al 2006).
2. Subjects with intermittent alcohol or substance use will not be excluded unless they have met DSM-IV criteria for current alcohol or substance dependence within the last 6 months or DSM-IV criteria for alcohol or substance abuse within the last month.
3. Subjects with nicotine use or dependence will not be excluded.
4. Subjects with daily marijuana use will be excluded because of the possibility of physical dependence on cannabis. Those with with marijuana use no more than once a week will not be excluded because such subjects will not be physically dependent on marijuana and so not at risk for rimonabant-elicited acute cannabis withdrawal. Experimental studies of human cannabis physical dependence and withdrawal suggest that high-dose, multiple times a day administration is needed to produce physical dependence (Jones et al., 1976; Haney et al., 1999)
5. Subjects with a history of Crohn's Disease or Irritable Bowel Syndrome
6. Subjects with a organic brain disorder
7. A DSM-IV eating disorder
8. Subjects with mental retardation will be excluded to exclude subjects with cognitive impairment not related to schizophrenia. Mental retardation will be determined by chart review for a mental retardation diagnosis or a history of an IQ <70 and functional disability noted before the age of 18 (DSM-IV criteria for mental retardation).
9. Subjects with a medical condition, whose pathology or treatment could alter the presentation or treatment of schizophrenia or significantly increase the risk associated with the proposed treatment protocol will be excluded.
10. Subjects with a history of surgical procedures for weight loss .
11. Subjects who are currently in the process of trying to quit cigarette smoking will be excluded.
12. Female subjects of childbearing potential must agree to use medically accepted means of contraception. Pregnant and lactating female subjects will be excluded. People with a diagnosis of diabetes will only be included if their diabetes is currently treated and under control and have been on their current medication regimen for at 3 months.
13. People with a blood pressure reading of 165/95 or greater at baseline will be excluded from the study.
14. The concomitant use of medications that are known to alter weight or appetite, including anti-obesity drugs; corticosteroids; or nicotine substitutes will not be allowed (see Appendix 2: Medication Exclusion List). 15. Additionally, patients treated with a form of valproate will not be included in the study.

16. Subjects must be judged competent to participate in the informed consent process (by passing the ESC with a score of 10/12) and provide voluntary informed consent.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2007-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Buchanan, MD, Principal Investigator — University of Maryland, College Park
Locations (4):
- United States (4):
  - Baltimore VA Medical Center, Baltimore, Maryland
  - Keypoint Health System, Baltimore, Maryland
  - Sheppard Pratt Health System, Baltimore, Maryland
  - Maryland Psychiatric Research Center (MPRC) Outpatient Research Program (ORP); the MPRC Treatment Research Program (TRP), Catonsville, Maryland

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 18 participants signed consent for the study. 1 participant was withdrawn prior to randomization, 2 participants (one from each group) withdrawn after randomization but prior to drug initiation. n=15 participants included in data analysis for aims 1, 2, 8, 9, 10, and n=14 analyzed for aims 3-7 due withdrawal prior to EOS neruopsych testing.
Groups:
- Rimonabant: Rimonabant: Rimonabant, 1 20 mg tablet given 1 time per day for 112 days.
- Placebo: Placebo
  Placebo: Placebo
Period: Overall Study
Arm/Group | Rimonabant | Placebo
Started | 8 | 9
Completed | 0 | 0
Not Completed | 8 | 9
Not completed — Did not qualify prior to starting drug | 1 | 1
Not completed — Study suspended | 7 | 8

BASELINE CHARACTERISTICS:
Population: 18 participants signed consent, 1 withdrawn prior to randomization, 17 subjects were randomized to study medication (rimonabant n=8, placebo n=9). Of these 17, 1 participant from each group was withdrawn prior to the receipt of study medication, thus n=15 analyzed for aims 1, 2,8,9,10; n=14 analyzed for aims 3-7.
Groups:
- Rimonabant: Rimonabant
  Rimonabant: Rimonabant, 1 20 mg tablet given 1 time per day for 112 days.
- Total: Total of all reporting groups
Arm/Group | Rimonabant | Placebo | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 15
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.9 (6.9) | 42.4 (13.3) | 45.7 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Brief Psychiatric Rating Scale (BPRS) Total Score
Description: The total BPRS score is calculated by adding the scores for scales #1-#18. Each scale ranges from "1=Not Present" to "7=Very Severe". Total scores range from a minimum score of 18 to a maximum score of 126. A higher total score indicates a more severe psychiatric symptom rating.
Time Frame: Baseline (Week 0) and end of study (Week 16)
Population: Because of early study termination, 2 participants on rimonabant and 3 on placebo were withdrawn before completion.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Placebo tablet given 1 time per day for 112 days
Arm/Group | Rimonabant | Placebo
Number analyzed (Participants) | 7 | 8
units on a scale
  Week 0 | 33.5 (7.5) | 34.5 (4.6)
  Week 16: number analyzed (Participants) | 5 | 5
  Week 16 | 32.8 (3.9) | 33.6 (6.2)

2. Primary Outcome: Brief Psychiatric Rating Scale (BPRS) Psychosis Score
Description: The psychosis score is calculated by adding the scores for scales #4 Conceptual Disorganization, #11 Suspiciousness, #12 Hallucinatory Behavior, and #15 Unusual Thought Content. Each scale ranges from "1=Not Present" to "7=Very Severe". The minimum psychosis score is 4 and the maximum psychosis score is 28. A higher score indicates a more severe psychosis rating.
Time Frame: Baseline (Week 0) and end of study (Week 16)
Population: Because of early study termination, 2 participants on rimonabant and 3 on placebo were withdrawn before completion.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rimonabant | Placebo
Number analyzed (Participants) | 7 | 8
units on a scale
  Week 0 | 9.4 (4.3) | 11.4 (3.4)
  Week 16: number analyzed (Participants) | 5 | 5
  Week 16 | 7.6 (3.0) | 8.6 (3.4)

3. Primary Outcome: The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)
Description: The RBANS is a brief, individually administered test designed to evaluate neuropsychological status of adults, ages 20-89. The 12 subtests measure attention, language, visuospatial/constructional abilities, and immediate and delayed memory. The raw scores from the subtests are scaled together to create index scores, and these are summed for conversion to a total scale score. Higher score equals a better outcome. The total index score range for the RBANS is 40-160.
Time Frame: Baseline (Week 0) and end of study (Week 16)
Population: 14 (R n=7, P n=7) completed baseline and End Of Study (EOS), 16 wk. Neurocognitive assessments (i.e. RBANS); 1 P pt. failed to complete the other EOS neurocognitive tests. 5 R pts. and 4 P pts. completed the 16-wk. treatment phase; the other 2 R pts. completed 11 and 13 wks. and 3 P pts. completed 13 (n=2) and 15 wks. (n=1).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rimonabant | Placebo
Number analyzed (Participants) | 7 | 7
units on a scale
  Week 0 | 85.0 (19.8) | 78.3 (10.2)
  Week 16 | 83.0 (11.8) | 84.3 (12.6)

4. Primary Outcome: The Iowa Gambling Task (IGT)
Description: The Iowa Gambling Task (IGT) is a computer-administered cognitive test that assesses risk preferences by simulating real-life decision making using uncertainty, rewards, and penalties. In the task, players are given four decks of cards and an endowment of fake money (e.g., $2000). Players are instructed to select cards one at a time and try to lose the least amount of money and win the most. The outcome measure was the number of rewarded minus punished card choices. Task has a maximum of 100 trials. The net score is the difference between the number of choices from advantageous decks verses disadvantageous decks. Higher scores are better and can range from -50 to +50.
Time Frame: Baseline (Week 0) and end of study (Week 16)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rimonabant | Placebo
Number analyzed (Participants) | 7 | 7
units on a scale
  Week 0 | 5.1 (19.8) | 1.3 (22.7)
  Week 16 | -0.3 (25.2) | -9.0 (29.7)

5. Primary Outcome: N-Back Neurocognitive Task: 0-back Condition
Description: The N-Back task is a sequential letter working memory task. D-prime was used to measure accuracy on the 0-back, 1-back, and 2-back conditions. D-prime scores range from 0 to 8.6. Higher scores are better. As memory load increases from 0 to 1, from 1 to 2, D-prime scores are expected to be lower.
Time Frame: Baseline (Week 0) and end of study (Week 16)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rimonabant | Placebo
Number analyzed (Participants) | 7 | 7
units on a scale
  Week 0 | 3.8 (0.5) | 3.6 (0.6)
  Week 16 | 3.9 (0.6) | 3.6 (0.4)

6. Primary Outcome: N-Back Neurocognitive Task: 1-back Condition
Description: as for outcome 5
Time Frame: Baseline (Week 0) and end of study (Week 16)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rimonabant | Placebo
Number analyzed (Participants) | 7 | 7
units on a scale
  Week 0 | 3.2 (0.8) | 3.2 (0.6)
  Week 16 | 3.3 (0.7) | 2.8 (0.2)

7. Primary Outcome: N-Back Neurocognitive Task: 2-back Condition
Description: as for outcome 5
Time Frame: Baseline (Week 0) and end of study (Week 16)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rimonabant | Placebo
Number analyzed (Participants) | 7 | 7
units on a scale
  Week 0 | 1.5 (0.6) | 1.6 (0.6)
  Week 16 | 1.5 (0.4) | 1.6 (0.4)

8. Secondary Outcome: Schedule for Assessment of Negative Symptoms (SANS) Total Score
Description: SANS total score range = 0-85. Higher scores indicate more severe negative symptoms.
Time Frame: Baseline (Week 0) and end of study (Week 16)
Population: Because of early study termination, 2 participants on rimonabant and 3 on placebo were withdrawn before completion.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rimonabant | Placebo
Number analyzed (Participants) | 7 | 8
units on a scale
  Week 0 | 28.7 (10.9) | 26.7 (15.5)
  Week 16: number analyzed (Participants) | 5 | 5
  Week 16 | 33.2 (11.6) | 32.4 (15.8)

9. Secondary Outcome: Schedule for Assessment of Negative Symptoms (SANS) - Anhedonia
Description: SANS Global Anhedonia score. Scores can range from 0-5, with higher scores indicating more severe anhedonia.
Time Frame: Baseline (Week 0) and end of study (Week 16)
Population: Because of early study termination, 2 participants on rimonabant and 3 on placebo were withdrawn before completion.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rimonabant | Placebo
Number analyzed (Participants) | 7 | 8
units on a scale
  Week 0 | 1.9 (1.0) | 1.6 (0.9)
  Week 16: number analyzed (Participants) | 5 | 5
  Week 16 | 1.9 (1.0) | 1.9 (1.1)

10. Secondary Outcome: Schedule for Assessment of Negative Symptoms (SANS) - Blunted Affect
Description: SANS Global Rating of Affective Flattening. Scores can range from 0-5, with higher scores indicating more severe blunted affect.
Time Frame: Baseline (Week 0) and end of study (Week 16)
Population: Because of early study termination, 2 participants on rimonabant and 3 on placebo were withdrawn before completion.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rimonabant | Placebo
Number analyzed (Participants) | 7 | 8
units on a scale
  Week 0 | 1.3 (0.9) | 1.1 (1.0)
  Week 16: number analyzed (Participants) | 5 | 5
  Week 16 | 1.8 (0.9) | 1.2 (1.0)

11. Secondary Outcome: Schedule for Assessment of Negative Symptoms (SANS) - Alogia
Description: SANS Global Rating of Alogia. Scores can range from 0-5, with higher scores indicating more severe alogia.
Time Frame: Baseline (Week 0) and end of study (Week 16)
Population: Because of early study termination, 2 participants on rimonabant and 3 on placebo were withdrawn before completion.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rimonabant | Placebo
Number analyzed (Participants) | 7 | 8
units on a scale
  Week 0 | 0.5 (0.5) | 0.9 (1.4)
  Week 16: number analyzed (Participants) | 5 | 5
  Week 16 | 0.9 (1.1) | 1.4 (1.3)

12. Secondary Outcome: Schedule for Assessment of Negative Symptoms (SANS) - Avolition
Description: SANS Avolition score. Scores can range from 0-5, with higher scores indicating more severe avolition.
Time Frame: Baseline (Week 0) and end of study (Week 16)
Population: Because of early study termination, 2 participants on rimonabant and 3 on placebo were withdrawn before completion.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rimonabant | Placebo
Number analyzed (Participants) | 7 | 8
units on a scale
  Week 0 | 2.6 (1.1) | 2.4 (1.1)
  Week 16: number analyzed (Participants) | 5 | 5
  Week 16 | 2.6 (1.2) | 3.0 (1.2)

13. Secondary Outcome: Clinical Global Impression (CGI)
Description: The global improvement score can range from 1-7, with higher scores indicating worse total improvement clinically.
Time Frame: Baseline (Week 0) and end of study (Week 16)
Population: Because of early study termination, 2 participants on rimonabant and 3 on placebo were withdrawn before completion.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rimonabant | Placebo
Number analyzed (Participants) | 7 | 8
units on a scale
  Week 0 | 4.2 (0.4) | 4.2 (0.7)
  Week 16: number analyzed (Participants) | 5 | 5
  Week 16 | 4.2 (0.4) | 4.0 (1.0)

14. Secondary Outcome: Calgary Depression Scale (CDS) Total Score
Description: The CDS total score is the addition of scores from items 1-9. Each item's scores range on a scale of "0=Absent" to "3=Severe". The total score range is from 0-27. Higher total scores indicate a more severe depression rating.
Time Frame: Baseline (Week 0) and end of study (Week 16)
Population: Because of early study termination, 2 participants on rimonabant and 3 on placebo were withdrawn before completion.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rimonabant | Placebo
Number analyzed (Participants) | 7 | 8
units on a scale
  Week 0 | 3.0 (2.2) | 3.0 (2.4)
  Week 16: number analyzed (Participants) | 5 | 5
  Week 16 | 2.0 (2.5) | 2.0 (2.7)

ADVERSE EVENTS:
Time Frame: Adverse effects identified by standard querying for new onset or worsened symptoms on a standard checklist administered bi-weekly.
Description: Side Effect Check (SEC) List was used
Arm/Group | Rimonabant | Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 4/8 | 6/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rimonabant (N=8) | Placebo (N=9)
Headache (General disorders) | 3 | 5
Enuresis (Renal and urinary disorders) | 3 | 4
Anorexia (Metabolism and nutrition disorders) | 3 | 3
Sedation (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Abdominal pain (Gastrointestinal disorders) | 3 | 4
weight loss (Metabolism and nutrition disorders) | 2 | 4
malaise (General disorders) | 2 | 3
tinnitus (Ear and labyrinth disorders) | 3 | 2
nausea (Gastrointestinal disorders) | 2 | 2
dizziness (General disorders) | 2 | 2
dry mouth (General disorders) | 2 | 2
insomnia (General disorders) | 1 | 3
vomiting (General disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes